CLINICAL TRIAL: NCT00869492
Title: A Double Blind Randomised Comparison of Nadifloxacin 1% Cream Alone and Nadifloxacine %1 Cream With Benzoyl Peroxide 5% Solution in the Treatment of Mild to Moderate Facial Acne Vulgaris
Brief Title: Comparison of Nadifloxacin Cream Alone and With Benzoyl Peroxide Solution in the Treatment of Acne
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Züleyha Yazıcı, Dermatology Department of Marmara University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mar-der1; dermatology1
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Acne Vulgaris
Keywords: Acne; Nadifloxacin; benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): instructed nadifloxacine 1% cream twice dailly, and placebo for benzoyl peroxide 5% solution once dailly
  Interventions: Drug: nadifloxacine
- B (Other): instructed nadifloxacine 1% cream twice dailly, and active benzoyl peroxide 5% solution once dailly
  Interventions: Drug: benzoyl peroxide; Drug: nadifloxacine

INTERVENTIONS:
Drug: benzoyl peroxide — benzoyl peroxide %5 solution once dailly
  Other Names: Aknefug BP5 lotion
  Arms: B
Drug: nadifloxacine — Nadifloxacine 1% cream twice dailly
  Other Names: Nadixa 1% cream

SUMMARY:
The purpose of this study is to determine whether using of nadifloxacine 1% cream and benzoyl peroxide 5% solution together is more effective than using nadifloxacine alone in the treatment of mild to moderate facial acne.

DETAILED DESCRIPTION:
Nadifloxacin; a new topical antibiotic for the treatment of acne has recently been marketed in our country. Only a few studies on its use and effectiviness could be found in the literature. Nadifloxacin may be an alternative to other topical antibiotics and benzoyl peroxide or its use along with benzoyl peroxide may be more effective and rational to prevent possible future resistance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate facial acne vulgaris
* Must have at least 10 inflammatory and/or non-inflammatory and no more than 3 nodulocystic acne lesions

Exclusion Criteria:

* Nodulocystic acne lesions more than 3 and pure comedonal acne
* Additional truncal acne needs systemic therapy
* Usage of topical treatments for acne in last 2 weeks, systemic antibiotic in last 4 weeks, systemic isotretinoin in last 6 months
* Application of chemical peels and laser in last 4 weeks
* Usage of hormones in last 3 months
* Clinical signs of hyperandrogenism in females
* Pregrancy and lactation
* Hypersensitivity to interventions
* Additional facial skin diseases (eg. atopic and seborreic dermatitis)
* Photosensitive disorders and usage of drugs which can trigger Photosensitive conditions

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients whom inflammatory lesions were decreased %50 or more | two months

SECONDARY OUTCOMES:
the number of patients whom were observed side effects | two months

CONTACTS AND LOCATIONS:
Overall Officials: Züleyha Yazıcı, doktor, Principal Investigator — Marmara University
Locations (1):
- Marmara University school of medicine, Istanbul, Turkey (Türkiye)